CLINICAL TRIAL: NCT01564485
Title: Role of Cardiac CT in Risk Factor Control in Asymptomatic Patients With Diabetes
Brief Title: Cardiac CT's Role in Asymptomatic Patients With Diabetes and Metabolic Syndrome
Acronym: CTRAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Shaista Malik, Assistant Professor, University of California, Irvine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008-6170
Record Dates: First submitted 2012-02-24; First posted 2012-03-27 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome | interventions — Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cardiac CT (Experimental): Patients randomized to cardiac CT will obtain a non-invasive assessment of their coronary arteries.
  Interventions: Diagnostic Test: Cardiac CT
- Usual Care (Active Comparator): Patients randomized to usual care will be assigned to continuing usual medical care with their primary care physician
  Interventions: Behavioral: Usual medical care

INTERVENTIONS:
Diagnostic Test: Cardiac CT — A cardiac CT involves a non-invasive test of the coronary arteries.
  Arms: Cardiac CT
Behavioral: Usual medical care — Patients would be treated by their primary care physicians with usual medical care with drugs such as lipid lowering medication, blood pressure lowering medications, and blood glucose lowering medications. The study will not specify which drugs to use and will it up to the individual physician's discretion.
  Other Names: Usual medical care would include control of blood pressure, blood glucose, and cholesterol by the primary care physician.
  Arms: Usual Care

SUMMARY:
This study looked at the role of cardiac CT in improving risk factor control in those with diabetes.

DETAILED DESCRIPTION:
This study examined whether doing a cardiac screening test, the cardiac CT, would result in patients paying more attention to controlling their risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Diabetes
* Metabolic Syndrome

Exclusion Criteria:

* Symptoms of heart disease
* Heart Disease
* Renal disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2008-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaista Malik, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data is now available
Access Criteria: We will need written request to share data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiac CT | Usual Care
Started | 92 | 101
Completed | 84 | 78
Not Completed | 8 | 23

BASELINE CHARACTERISTICS:
Groups:
- Cardiac CT Group: Asymptomatic patients with Type II DM who received cardiac CT screening test
- Usual Care Group: Asymptomatic patients with Type II DM who received usual care
- Total: Total of all reporting groups
Arm/Group | Cardiac CT Group | Usual Care Group | Total
Number analyzed (Participants) | 92 | 101 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 91 | 176
  >=65 years | 7 | 10 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 58 | 112
  Male | 38 | 43 | 81

OUTCOME MEASURES:

1. Primary Outcome: Systolic BP Pressure
Description: After randomization to either obtain cardiac CT or usual care, patients will be followed for 5 years (with assessment of outcomes at every 6 months) to see any difference in control of systolic blood pressure. The outcome with be assessed as a continuous measure.
Time Frame: Five year follow up
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Cardiac CT | Usual Care
Number analyzed (Participants) | 75 | 72
mm Hg | 145 (6) | 144 (5)

2. Other Pre Specified Outcome: Change in Treatment by PCP
Description: Medication dose change or medication start/stop
Time Frame: 2 years
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change in Treatment by PCP
Description: Medication dose change or medication start/stop
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Description: No adverse events
Arm/Group | Cardiac CT | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/93
Other Adverse Events (participants affected / at risk) | 0/92 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No